CLINICAL TRIAL: NCT01866332
Title: Effectiveness of the Addition of the Kinesio Taping Method to Conventional Physical Therapy Treatment in Patients With Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of the Addition of the Kinesio Taping Method to Conventional Physical Therapy Treatment in Patients With Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciola da Cunha Menezes Costa, Associate Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAPESP2013/02075-8; 02075-8 (Other Grant/Funding Number: FAPESP, Brazil)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Nonspecific Chronic Low Back Pain
Keywords: back pain; tape; chronic
MeSH Terms: conditions — Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Musculoskeletal Manipulations; Exercise Therapy; Bandages; Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Physical Therapy (Active Comparator): Combination of manual therapy techniques, general exercises and specific exercises for spinal segmental stabilization. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week). The treatment will be tailored to the patient presentation (i.e. pragmatic treatment).
  Interventions: Other: Conventional Physical Therapy
- Conventional Physical Therapy plus Kinesiotaping (Experimental): Patients will receive conventional physical therapy plus an application of Kinesiotaping in their lumbar spine.
  Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week).
  Interventions: Other: Conventional Physical Therapy; Device: Kinesio Tex Gold ( Kinesiotaping )

INTERVENTIONS:
Other: Conventional Physical Therapy — Combination of manual therapy techniques, general exercises and specific exercises for spinal segmental stabilization. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week). The treatment will be tailored to the patient presentation (i.e. pragmatic treatment).
  Other Names: Manual therapy; Exercise therapy; Specific exercises
Device: Kinesio Tex Gold ( Kinesiotaping ) — Kinesiotaping intervention is based upon the use of specific elastic tapes (known as Kinesio Tex Gold) that are applied with a certain amount of tension fixed to the skin of patients with the target muscles in a stretched position. The tapes will be placed over the superficial back muscles (erector spinae muscles).
  Other Names: Bandages; Tape; Taping; Kinesio Tex; Kinesio Tape; Kinesiotape
  Arms: Conventional Physical Therapy plus Kinesiotaping

SUMMARY:
The purpose of this study is to determine the effectiveness of the addition of the use of Kinesio Taping in patients with chronic nonspecific low back pain who receive conventional physical therapy.

DETAILED DESCRIPTION:
One hundred and forty-eight patients will be randomized to receive either conventional physical therapy, which consist of a combination of manual therapy techniques, general exercises and specific exercises for spinal segmental stabilization (Conventional Physical Therapy Group) or to receive conventional physical therapy plus the addition of the Kinesio Taping in the lumbar spine (Conventional Physical Therapy plus Kinesio Taping), over a period of 5 weeks (10 sessions of treatment).

Clinical outcomes (pain intensity, disability and global perceived effect ) will be collected at baseline and at 5 weeks, 3 and 6 months after randomization. Data will be collected by a blinded examiner who will be unaware about the group allocation. All statistical analysis will be conducted following the principles of intention to treat analysis and the between-group differences will be performed using Mixed Linear Models.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific low back pain longer than 12 weeks
* Seeking care for low back pain

Exclusion Criteria:

* Contra indications to physical exercise
* Serious spinal pathologies (e.g. tumors, fractures and inflammatory diseases)
* Nerve root compromise
* Contra indications to the Kinesio Taping (e.g. intolerance to tapes, band aids etc)
* Pregnancy
* Severe cardiorespiratory conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Five weeks after randomization
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability | Five weeks after randomization
  Disability associated with low back pain will be measured by the 24-item Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Pain Intensity | 3 and 6 months after randomization
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability | 3 and 6 months after randomization
  Disability associated with low back pain will be measured by the 24-item Roland Morris Disability Questionnaire
Global impression of recovery | 5 weeks, 3 and 6 months after randomization
  Global impression of recovery will be measured by an 11-point (-5 to +5) Global Perceived Effect Scale

OTHER OUTCOMES:
Satisfaction with care | 5 weeks after randomization
  Satisfaction with care will be measured by the Medrisk Instrument for Measuring Patient Satisfaction with Physiotherapy Care

CONTACTS AND LOCATIONS:
Overall Officials: Luciola CM Costa, PhD, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Physical Therapy Outpatient Department, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Added MA, Costa LO, de Freitas DG, Fukuda TY, Monteiro RL, Salomao EC, de Medeiros FC, Costa Lda C. Kinesio Taping Does Not Provide Additional Benefits in Patients With Chronic Low Back Pain Who Receive Exercise and Manual Therapy: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2016 Jul;46(7):506-13. doi: 10.2519/jospt.2016.6590. Epub 2016 Jun 6. PMID 27266883
- See also: Info from the grant sponsor of this study (FAPESP, Brazil) — http://www.bv.fapesp.br/pt/pesquisador/665136/luciola-da-cunha-menezes-costa/